CLINICAL TRIAL: NCT05673174
Title: Assessment of the Vivio System for the Non-Invasive Estimation of Left Ventricular Diastolic Pressure (LVDP) in Healthy Volunteers
Brief Title: Avicena LVDP Validation Study in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Avicena LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-0006
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: left ventricular diastolic pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Non-Invasive Estimation of Left Ventricular Diastolic Pressure — Modified blood pressure cuff used to detect arterial waveforms used for the estimation of LVDP

SUMMARY:
The purpose of this study is to document the utility of the Vivio System in quantifying LVDP in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects >21 years of age.
2. No known significant health problems.
3. Willing and able to participate in all study evaluations.
4. Ability to understand and sign informed consent.

Exclusion Criteria:

1. Open skin lesions at the site of Vivio application / examination.
2. Inability to obtain brachial artery blood pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers, no history of Heart Disease.
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
To construct an algorithm from training data set to be used to estimate the ROC curve from the algorithm for a separate test data set. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Avicena, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: Undecided